CLINICAL TRIAL: NCT01686555
Title: Assessment of the Safety, Tolerability, and Pharmacokinetics of ABT-199 After Single and Multiple Ascending Doses in Female Subjects With Systemic Lupus Erythematosus (SLE)
Brief Title: A Study to Evaluate the Safety, Tolerability and Pharmacokinetics of ABT-199 in Female Patients With Systemic Lupus Erythematosus (SLE)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: M13-093; 2013-000328-33 (EudraCT Number)
Record Dates: First submitted 2012-09-13; First posted 2012-09-18 (Estimated); Last update posted 2017-11-20 (Actual); Status verified 2015-07

CONDITIONS: Lupus Erythematosus
MeSH Terms: interventions — venetoclax

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Single Dose (Experimental): Subjects enrolled in the Single Ascending Dose (SAD) part of the study will receive a single dose of study drug or placebo. (Groups 1, 2, 3, 4, 5 and 6).
  Interventions: Drug: ABT-199; Other: Placebo
- Multiple Dose (Experimental): Subjects enrolled in the Multiple Ascending Dose (MAD) part of the study will receive multiple doses of study drug or placebo. (Groups 7, 8, 9, 10 and 11)
  Interventions: Drug: ABT-199; Other: Placebo

INTERVENTIONS:
Drug: ABT-199 — Tablet
Other: Placebo — Tablet

SUMMARY:
To assess the safety, tolerability and pharmacokinetics of ABT-199 in female subjects with Systemic Lupus Erythematosus.

DETAILED DESCRIPTION:
This is a phase 1, randomized, double-blind, placebo-controlled, single-and multiple ascending dose study. Up to eighty-eight subjects with Systemic Lupus Erythematosus will be selected to participate. Subjects will be randomized to receive either ABT-199 or placebo. Subjects will be administered ABT-199/placebo as a single dose or up to 14 days as multiple doses.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of systemic lupus erythematosus for at least 6 months.
* Documentation of at least one of the following: ANA titer >= 1:160 or positive anti-dsDNA antibodies.
* Stable systemic lupus erythematosus medication regimen.
* Other than systemic lupus erythematosus, subject should be in general good health.

Exclusion Criteria:

* Male.
* Drug-induced or highly active systemic lupus erythematosus.
* Significant autoimmune disease other than lupus.
* Significant, uncontrolled or unstable disease in any organ.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2012-11; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Number of participants with Adverse Events | From first dose of ABT-199 until 28 days after single dose of ABT-199 and until 21 days after the last multiple dose of ABT-199
  Collect all adverse events at each visit
Physical Exam including vital signs | Prior to the first dose of ABT-199 until 28 days after single dose of ABT-199 and until 21 days after the last multiple dose of ABT-199
  Blood pressure, heart rate and body temperature
Clinical Lab Testing | Prior to the first dose of ABT-199 until 28 days after single dose of ABT-199 and until 21 days after the last multiple dose of ABT-199
  Hematology, Chemistry, and Urinalysis
Electrocardiogram (ECG) Measurements | For 24 hours after a single dose of ABT-199 and up to 24 hours after the seventh dose of multiple doses of ABT-199
  ECGs done in triplicate
Maximum observed serum concentration (Cmax) of ABT-199 | For 72 hours after a single dose of ABT-199 and for 24 hours after the seventh dose of multiple doses of ABT-199
  Cmax
Time to Cmax (Tmax) of ABT-199 | For 72 hours after a single dose of ABT-199 and for 24 hours after the seventh dose of multiple doses of ABT-199
  Time to Cmax
The area under the time curve (AUC) of ABT-199 | For 72 hours after a single dose of ABT-199 and for 24 hours after the seventh dose of multiple doses of ABT-199
  the area under the exposure-time curve of ABT-199 extrapolated to infinite time for single doses and up to 24 hrs for multiple doses of ABT-199
The terminal phase elimination rate constant and the terminal elimination half-life (t1/2) of ABT-199 | For 72 hours after a single dose of ABT-199
  The terminal phase elimination rate constant and the terminal elimination half-life (t1/2) of ABT-199

SECONDARY OUTCOMES:
Measurement of lymphocyte depletion and recovery | Prior to the first dose of ABT-199 until 28 days after single dose of ABT-199 and until 21 days after the last multiple dose of ABT-199
  explore pharmacokinetic/pharmacodynamic relationship

CONTACTS AND LOCATIONS:
Overall Officials: Peng Lu, MD, Study Director — AbbVie
Locations (15):
- United States (11):
  - Site Reference ID/Investigator# 89694, Clearwater, Florida
  - Site Reference ID/Investigator# 131720, DeBary, Florida
  - Site Reference ID/Investigator# 118637, Miami, Florida
  - Site Reference ID/Investigator# 124116, Miami Lakes, Florida
  - Site Reference ID/Investigator# 89693, Orlando, Florida
  - Site Reference ID/Investigator# 78256, Overland Park, Kansas
  - Site Reference ID/Investigator# 129826, Rochester, Minnesota
  - Site Reference ID/Investigator# 89773, Manhasset, New York
  - Site Reference ID/Investigator# 78254, Duncansville, Pennsylvania
  - Site Reference ID/Investigator# 123335, Dallas, Texas
  - Site Reference ID/Investigator# 78253, Dallas, Texas
- Site Reference ID/Investigator# 107896, Berlin, Germany
- Mexico (2):
  - Site Reference ID/Investigator# 116395, Distrito Federal
  - Site Reference ID/Investigator# 112555, Monterrey
- Site Reference ID/Investigator# 132009, San Juan, Puerto Rico

REFERENCES:
- [Result] Lu P, Fleischmann R, Curtis C, Ignatenko S, Clarke SH, Desai M, Wong SL, Grebe KM, Black K, Zeng J, Stolzenbach J, Medema JK. Safety and pharmacodynamics of venetoclax (ABT-199) in a randomized single and multiple ascending dose study in women with systemic lupus erythematosus. Lupus. 2018 Feb;27(2):290-302. doi: 10.1177/0961203317719334. Epub 2017 Jul 10. PMID 28691866
- [Derived] Nader A, Minocha M, Othman AA. Exposure-Response Analyses of the Effects of Venetoclax, a Selective BCL-2 Inhibitor, on B-Lymphocyte and Total Lymphocyte Counts in Women with Systemic Lupus Erythematosus. Clin Pharmacokinet. 2020 Mar;59(3):335-347. doi: 10.1007/s40262-019-00818-5. PMID 31541431
- [Derived] Minocha M, Zeng J, Medema JK, Othman AA. Pharmacokinetics of the B-Cell Lymphoma 2 (Bcl-2) Inhibitor Venetoclax in Female Subjects with Systemic Lupus Erythematosus. Clin Pharmacokinet. 2018 Sep;57(9):1185-1198. doi: 10.1007/s40262-017-0625-2. PMID 29333561